CLINICAL TRIAL: NCT04014894
Title: Safety and Efficiency Study of ET019003-T Cells in Relapsed/Refractory CD19+ B-Cell Leukemia and Lymphoma
Brief Title: ET019003-T Cells in Relapsed/Refractory CD19+ B-Cell Leukemia and Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Eureka(Beijing) Biotechnology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, MEI HENG, Principal Investigator, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET019003-T
Record Dates: First submitted 2019-07-02; First posted 2019-07-10 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Intervention Model Description: This study was a single-center, open-label, single-arm, non-randomized,3+3 dose escalation clinical trial.18 patients are separated into 9 leukemia and 9 lymphoma. Each disease has 3 groups by infusion dose level. Each dose group has 3 patients.If no DLT emerges in the group, then the next group uses the subsequent higher dose. If DLT emerges in a single subject in any dose level, 3 more subjects will be enrolled to the same dose level.The maximum dose could be extended.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ET019003-T Cells (Experimental): The trial will enroll 9 patients with leukemia and 9 patients with lymphoma. Each disease has 3 dose-levels.
  Interventions: Drug: ET019003-T Cells

INTERVENTIONS:
Drug: ET019003-T Cells — Fludarabine 25 mg/day on day -5, -4 and -3; Cyclophosphamide 250 or 300 mg/day on day -5, -4 and -3; ET019003-T Cells on day 0.

SUMMARY:
This is a single center, open-label, 3+3 dose escalation, phase 1 study to evaluate the efficacy and safety of ET019003-T cells therapy for patients with relapsed/refractory CD19+ acute lymphoblastic leukemia and lymphoma.

DETAILED DESCRIPTION:
ET019003-T cells is a human anti-CD19 CAR-T cells by fusing the anti-CD19 antibody Fab domain with the transmembrane and intracellular domains from the γδTCR, which can avoid mispairing with the T cell's endogenous αβTCR chains. Meanwhile, an independent ET190L1-CSR(Chimeric Signaling Receptor) is added to ET019003-T cells in trans, which can bind CD19 to activate a novel costimulatory domain to further promote T cell proliferation and persistence.

The trial is conducted to explore the safety and efficacy of ET019003-T cells in CD19+ Leukemia and Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or his or her legal guardian voluntarily participates in and signs an informed consent form.
2. Male or female, aged 18 to 75 years (including 18 and 75 years old).
3. Pathologically confirmed CD19+ B-cell malignancies, and patients met the following criteria for refractory or relapsed B-cell malignancies.

   A. Refractory/relapsed B-cell lymphoblastic leukemia (meeting one of the following) i. Recurrence within 6 months after first remission. ii. Primary refractory disease which cannot achieve complete remission (CR) after 2 cycles of standardized chemotherapy regimen.

   iii. Failure to achieve CR or relapse after one line or multiple lines of salvage chemotherapy.

   iv. Not suitable for hematopoietic stem cell transplantation (HSCT), or abandon HSCT due to various restrictions, or relapse after HSCT.

   B. Refractory/relapsed B-cell lymphoma (Meeting 1 of the first 3 items plus item 4) i. Tumor shrinkage less than 50% or disease progression after 4 cycles of standard chemotherapy.

   ii. Achieved CR after standard chemotherapy, but relapsed within 6 months. iii. Two or more relapses after CR. iv. Subjects must have received adequate treatment in the past, including anti-CD20 monoclonal antibody and combination chemotherapy with anthracyclines.
4. Having a measurable or evaluable lesion:

   A. Patients with lymphoma require a single lesion≥15mm or 2 or more lesions≥10mm.

   B. Patients with leukemia require persistent positive or positive relapse of bone marrow MRD.
5. Patient's main organs functioning well:

   A. Liver function: ALT/AST ≤ 3 times the upper limit of normal (ULN) and total bilirubin≤2 times ULN.

   B. Renal function: Creatinine < 220μmol/L. C. Pulmonary function: Indoor oxygen saturation≥95%. D. Cardiac Function: Left ventricular ejection fraction (LVEF) ≥ 50%.
6. ≥ 2 weeks since prior therapy at the time of enrollment, and the toxicity related to previous treatments returned to < grade 1 (except for low grade toxicity such as alopecia).
7. ECOG score≤ 2.
8. Estimated survival time≥3 months.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. Women of child-bearing potential and all male participants can't use effective methods of contraception for at least 12 months following infusion.
3. Patients fail to collect enough PBMC.
4. Patients with other uncontrolled diseases, such as active infections.
5. Active hepatitis B or active hepatitis C.
6. Known HIV positive patients.
7. Patients with active autoimmune diseases requiring systemic immunosuppressive therapy.
8. Participants with other active malignancies (except non-melanoma skin cancer and cervical cancer) within 3 years.
9. Patients with severe mental disorder or disorders of consciousness.
10. Patients who need immediate treatment to control tumor progression or relieve tumor burden.
11. Patients participated in other clinical treatments within 6 weeks.
12. Patients with drug addiction.
13. Patients with poor treatment compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2019-06-12 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | 3 years
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0).

SECONDARY OUTCOMES:
Overall Remission Rate(ORR) of ET019003-T cells in Leukemia and Lymphoma | 3 years
  ORR will be assessed from the first CAR-T cell infusion to death or last follow-up (censored).
Overall survival(OS) of ET019003-T cells in Leukemia and Lymphoma | 3 years
  OS will be assessed from the first CAR-T cell infusion to death or last follow-up (censored).
Progress-free survival(PFS) of ET019003-T cells in Leukemia and Lymphoma | 3 years
  PFS will be assessed from the first CAR-T cell infusion to death or last follow-up (censored).
duration of Response(DOR) of ET019003-T cells in Leukemia and Lymphoma | 3 years
  DOR will be assessed from the first CAR-T cell infusion to death or last follow-up (censored).
Rate of ET019003-T cells in bone marrow cells and peripheral blood cells | 3 years
  In vivo (bone marrow and peripheral blood) rate of ET019003-T cells were determined by means of flow cytometry.
Quantity of ET019003-T CAR copies in bone marrow cells and peripheral blood cells | 3 years
  In vivo (bone marrow and peripheral blood) quantity of ET019003-T CAR copies copies were determined by means of qPCR.

CONTACTS AND LOCATIONS:
Overall Officials: Heng Mei, M.D., Ph.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Background] Schuster SJ, Bishop MR, Tam CS, Waller EK, Borchmann P, McGuirk JP, Jager U, Jaglowski S, Andreadis C, Westin JR, Fleury I, Bachanova V, Foley SR, Ho PJ, Mielke S, Magenau JM, Holte H, Pantano S, Pacaud LB, Awasthi R, Chu J, Anak O, Salles G, Maziarz RT; JULIET Investigators. Tisagenlecleucel in Adult Relapsed or Refractory Diffuse Large B-Cell Lymphoma. N Engl J Med. 2019 Jan 3;380(1):45-56. doi: 10.1056/NEJMoa1804980. Epub 2018 Dec 1. PMID 30501490
- [Background] Maude SL, Laetsch TW, Buechner J, Rives S, Boyer M, Bittencourt H, Bader P, Verneris MR, Stefanski HE, Myers GD, Qayed M, De Moerloose B, Hiramatsu H, Schlis K, Davis KL, Martin PL, Nemecek ER, Yanik GA, Peters C, Baruchel A, Boissel N, Mechinaud F, Balduzzi A, Krueger J, June CH, Levine BL, Wood P, Taran T, Leung M, Mueller KT, Zhang Y, Sen K, Lebwohl D, Pulsipher MA, Grupp SA. Tisagenlecleucel in Children and Young Adults with B-Cell Lymphoblastic Leukemia. N Engl J Med. 2018 Feb 1;378(5):439-448. doi: 10.1056/NEJMoa1709866. PMID 29385370
- [Background] Neelapu SS, Locke FL, Bartlett NL, Lekakis LJ, Miklos DB, Jacobson CA, Braunschweig I, Oluwole OO, Siddiqi T, Lin Y, Timmerman JM, Stiff PJ, Friedberg JW, Flinn IW, Goy A, Hill BT, Smith MR, Deol A, Farooq U, McSweeney P, Munoz J, Avivi I, Castro JE, Westin JR, Chavez JC, Ghobadi A, Komanduri KV, Levy R, Jacobsen ED, Witzig TE, Reagan P, Bot A, Rossi J, Navale L, Jiang Y, Aycock J, Elias M, Chang D, Wiezorek J, Go WY. Axicabtagene Ciloleucel CAR T-Cell Therapy in Refractory Large B-Cell Lymphoma. N Engl J Med. 2017 Dec 28;377(26):2531-2544. doi: 10.1056/NEJMoa1707447. Epub 2017 Dec 10. PMID 29226797
- [Background] Xu Y, Yang Z, Horan LH, Zhang P, Liu L, Zimdahl B, Green S, Lu J, Morales JF, Barrett DM, Grupp SA, Chan VW, Liu H, Liu C. A novel antibody-TCR (AbTCR) platform combines Fab-based antigen recognition with gamma/delta-TCR signaling to facilitate T-cell cytotoxicity with low cytokine release. Cell Discov. 2018 Nov 20;4:62. doi: 10.1038/s41421-018-0066-6. eCollection 2018. PMID 30479831
- [Derived] Li C, Zhou F, Wang J, Chang Q, Du M, Luo W, Zhang Y, Xu J, Tang L, Jiang H, Liu L, Kou H, Lu C, Liao D, Wu J, Wei Q, Ke S, Deng J, Liu C, Mei H, Hu Y. Novel CD19-specific gamma/delta TCR-T cells in relapsed or refractory diffuse large B-cell lymphoma. J Hematol Oncol. 2023 Jan 21;16(1):5. doi: 10.1186/s13045-023-01402-y. PMID 36681817